CLINICAL TRIAL: NCT04498923
Title: Duration of Blockade of Peripheral Nerves With Low Concentrated Bupivacaine Solution Depending of the Adjuvants
Brief Title: Duration of Blockade of Peripheral Nerves With Bupivacaine Depending of the Adjuvants
Acronym: DBBA
Status: Completed | Type: Observational
Sponsor: Lviv National Medical University (Other)
Responsible Party: Principal Investigator, Maksym Barsa, Principal Investigator, Lviv National Medical University
Other Study IDs: LNMY-FPGE- ANESTHESIOLOGY-DBBA
Record Dates: First submitted 2020-07-29; First posted 2020-08-05 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-04

CONDITIONS: Postoperative Pain; Peripheral Neuropathy; Fractures of the Upper Limb; Fracture of the Lower Limb (Except Hip), Initial Encounter; Intraoperative Hypotension; Intraoperative Hypertension; Pain Syndrome; Anesthesia; Anesthesia, Local; Local Anesthetic Systemic Toxicity
Keywords: Regional anesthesia; Pain management; Local anesthetic; Electromyography
MeSH Terms: conditions — Pain, Postoperative; Peripheral Nervous System Diseases; Somatoform Disorders; Agnosia | interventions — Bupivacaine; Dexamethasone; Epinephrine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Bupivacaine with dexamethasone: Ultrasound guided peripheral nerve block for upper or lower extremity was performed before orthopedic surgery using neurostimulator.
  Twenty milliliters solution of bupivacaine 0,375% with dexamethasone was injected for one plexus or peripheral nerve.
  Interventions: Drug: Bupivacaine, dexamethasone, epinephrine
- Bupivacaine with dexamethasone and epinephrine: Ultrasound guided peripheral nerve block for upper or lower extremity was performed before orthopedic surgery using neurostimulator.
  Twenty milliliters solution of bupivacaine 0,375% with dexamethasone 0,02% and epinephrine 0,00018% was injected for one plexus or peripheral nerve.
  Interventions: Drug: Bupivacaine, dexamethasone, epinephrine

INTERVENTIONS:
Drug: Bupivacaine, dexamethasone, epinephrine — Bupivacaine 75 mg, dexamethasone 4 mg, epinephrine 0,18 mg

SUMMARY:
The main aim of the investigator's study is to propose combination of local anesthetics and adjuvants that provides both adequate anesthesia during surgery and prolonged post-operative analgesia.

DETAILED DESCRIPTION:
Peripheral nerve plexuses blocks are performing as a component of analgesia in patients undergoing orthopedic surgery on the upper or lower extremities. Patients are divided into two groups depending on the adjuvant to the local anesthetic: 1st group - patients whose blockade is performed with a solution of bupivacaine 0.375% together with dexamethasone 0.02%; Group 2 - patients whose blockade is performed with a solution of bupivacaine 0.375% together with dexamethasone 0.02% and epinephrine 0.00018%. The duration of the blockade is estimated by puncturing the skin with a needle. The intensity of pain is assessed at 6, 12, 24 and 36 hours after blockade using Visual analog scale (VAS). The amount of narcotic anesthetic used in the postoperative period is also recorded. In addition, patients underwent electromyography of the innervation area of the blocked nerve before the surgery and 24 and 36 hours after surgery.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing upper or lower extremity orthopedic surgery

Exclusion Criteria:

* diabetes mellitus;
* diseases of the peripheral nerv system

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients undergoing orthopedic surgery on the upper and lower extremities in the Regional Center of Orthopedics, Traumatology and Vertebrology of Rivne Oblast State Hospital
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2022-04-05 (Actual); Study Completion 2022-04-05 (Actual)

PRIMARY OUTCOMES:
The duration of blockade | 6th, 12th, 24th and 36th hours after blockade
  The duration of the blockade was estimated by puncturing the skin with a needle every hour. In addition, patients underwent electromyography of the innervation area of the blocked nerve before the surgery and 24 and 36 hours after surgery.

SECONDARY OUTCOMES:
The amount of narcotic anesthetic used in the postoperative period | 48 hour after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Maksym Barsa, Principal Investigator — Сlinical resident
Locations (1):
- Rivne Oblast State Hospital, Rivne, Rivne Oblast, Ukraine

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: ORCID — https://orcid.org/0000-0002-2578-4935